CLINICAL TRIAL: NCT02270580
Title: Patient Navigation to Improve Quality of Life and Screening Practices Among Latino Breast Cancer Survivors
Brief Title: Komen Breast Cancer Survivor Health Screening Promotion Project: Staying Healthy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC20120059H
Record Dates: First submitted 2014-10-16; First posted 2014-10-21 (Estimated); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PN+ (Experimental): we will evaluate the efficacy of a culturally tailored PN program ("PN+") on improving quality of life (QoL), screening practices and treatment follow-up compliance among breast HL survivors
  Interventions: Behavioral: PN+
- PN usual (Active Comparator): participants will receive information brochures on breast cancer survivorship and have a minimum of 1 contact with the patient navigator
  Interventions: Behavioral: PN usual

INTERVENTIONS:
Behavioral: PN+ — we will evaluate the efficacy of a culturally tailored PN program ("PN+") on improving quality of life (QoL), screening practices and treatment follow-up compliance among breast HL survivors
  Arms: PN+
Behavioral: PN usual — participants will receive information brochures on breast cancer survivorship and have a minimum of 1 contact with the patient navigator
  Arms: PN usual

SUMMARY:
A randomized controlled trial (RCT) with 2 patient navigator conditions: PN+ and usual PN in which (condition 1) we will evaluate the efficacy of a culturally tailored PN program ("PN+") on improving quality of life (QoL), screening practices and treatment follow-up compliance among breast HL survivors. In usual PN, participants will receive information brochures on breast cancer survivorship and have a minimum of 1 contact with the patient navigator.

DETAILED DESCRIPTION:
This RCT involves a 2 (group) by 2 (time) repeated measures design with experimental condition (specialized PN+cancer survivorship program over 6 months versus PN only (control condition) as the between-groups factor, and time-point (baseline pre-randomization and post-PN at 6 months follow-up) as the within-groups factor. This RCT involves 2 patient navigator conditions: PN+ and usual PN in which (condition 1) we will evaluate the efficacy of a culturally tailored PN program ("PN+") on improving quality of life (QoL), screening practices and treatment follow-up compliance among breast HL survivors. In usual PN, participants will receive information brochures on breast cancer survivorship and have a minimum of 1 contact with the patient navigator.

ELIGIBILITY:
Inclusion Criteria:

* report a primary diagnosis of breast cancer
* have completed primary treatment within the past 36 months
* evidence of verbal fluency in English or Spanish
* self-identify as HL

Exclusion Criteria

* evidence of metastatic disease
* current severe mental illness such as psychosis
* substance dependence within the past year
* active suicidality
* ongoing neo-adjuvant therapy
* unavailable for follow-up over the course of the study period

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
General quality of life | 6 months
  The Functional Assessment of Cancer Therapy-General (FACT-G) will be administered to evaluate general domains of QOL. The FACT-G, now in its fourth revision, is one of the most widely used instruments to assess overall adjustment to cancer treatment and survivorship. It is a 27-item self-report questionnaire that takes less than 15 minutes to administer. The FACT-G assesses QOL in four domains of well-being: physical, social/family, emotional and functional well-being. Patients are asked to indicate the extent to which they agree with statements such as "I have pain," "I feel ill," "I get emotional support from my family," "I get support from my friends," "I feel sad," "I feel nervous," "I am sleeping well," and "I am content with the quality of my life right now." The scale is validated for use in many settings with many age groups. We will calculate a composite score for general QOL as well as subscale scores for specific domains of QOL.
Disease-specific quality of life | 6 months
  We will administer a cancer-specific FACT version, the FACT-B (breast cancer survivors). It addresses QOL issues that are common sequelae of that certain cancer.
Treatment follow-up compliance | 6 months
  Because all of our HL cancer survivors will be recruited within 12-months post-treatment completion for a primary tumor, we will follow ACS guidelines for follow-up care for one- to two-years post-treatment. We will assess via self-report whether the participant missed a scheduled follow-up appointment during the study period. A compliance categorical outcome measure (compliant vs. non-compliant) will be calculated for each participant. Compliance will be defined as attending all scheduled follow-up appointments specific to cancer treatment follow-up during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G Ramirez, DRPH, Principal Investigator — The University of Texas Health Science Center at San Antonio